CLINICAL TRIAL: NCT05285384
Title: An Open-Label, Single-Arm Clinical Trial to Evaluate the Immunogenicity and Safety of a Booster Dose of an Adjuvanted Recombinant Spike Protein COVID-19 Vaccine (SpikoGen) in Kidney Transplant Recipients After Two Doses of Sinopharm COVID-19 Vaccine
Brief Title: Immunogenicity and Safety of a Booster Dose of the SpikoGen Vaccine in Kidney Transplant Recipients After Two Doses of Sinopharm Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cinnagen (Industry)
Collaborators: Shahid Beheshti University of Medical Sciences (Other); Vaxine Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAC.CIN.PT.BOOSTER.KTR; IRCT20150303021315N28 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-COV-2; Recombinant protein; Spike; Advax-SM; Advax; Vaccine; Adjuvant; Kidney Transplant
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SpikoGen COVID-19 Vaccine (Experimental)
  Interventions: Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant

INTERVENTIONS:
Biological: SARS-CoV-2 recombinant spike protein + Advax-SM adjuvant — SARS-CoV-2 recombinant spike protein (25 μg) with Advax-SM adjuvant (15 mg); a single intramuscular injection into the deltoid muscle of the non-dominant arm
  Other Names: SpikoGen; COVAX-19

SUMMARY:
This is an open-label, single-arm clinical trial designed to evaluate the immunogenicity and safety of a booster dose of an adjuvanted recombinant SARS-CoV-2 spike protein subunit vaccine (SpikoGen) produced by CinnaGen Co. in kidney transplant recipients after two doses of Sinopharm's inactivated virus vaccine. A total of 100 adult individuals receive a single dose of the SpikoGen COVID-19 vaccine at 1 to 3 months after the second dose of the Sinopharm COVID-19 vaccine. The injection is given in the deltoid muscle of the non-dominant arm. For immunogenicity assessments, blood samples will be collected one month after the booster injection. For safety assessments, all participants will be followed up for one month.

Study hypotheses include:

1. A booster dose of the SpikoGen COVID-19 vaccine induces strong immunogenicity against SARS-CoV-2 in adult kidney transplant recipients who were fully vaccinated with Sinopharm COVID-19 vaccine.
2. A booster dose of the SpikoGen COVID-19 vaccine is safe and tolerable in adult kidney transplant recipients who were fully vaccinated with Sinopharm COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years
* Willing and able to comply with all study requirements, including scheduled visits, intervention, and laboratory tests
* Kidney transplant recipients who had received two doses of Sinopharm vaccine after transplantation
* Females must not be pregnant or breastfeeding
* At least six months should have passed from the time of transplantation
* Between 1 to 3 months should have passed from the second dose of Sinopharm vaccine

Exclusion Criteria:

* Subjects with signs of active SARS-CoV-2 infection at the screening visit
* Subjects with a history of SARS-CoV-2 infection based on a positive PCR test result after the second dose of the primary vaccination
* Subjects with an active CMV infection that requires treatment
* Subjects who have received rituximab within 6 months prior to the screening visit
* Subjects who have received intravenous immune globulin (IVIG) within 6 months prior to the screening visit
* Subjects who have a history of severe allergic reactions (e.g., anaphylaxis) to the study vaccine, any components of the study interventions, or any pharmaceutical products.
* Subjects who have received any other investigational products within 30 days prior to the screening visit or intend to participate in any other clinical studies during the period of this study.
* Subjects who have experienced transplant rejection within 30 days prior to the screening visit
* Subjects with any condition that may increase the risk of participating in the study or may interfere with the evaluation of the primary endpoints of the study in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with seroconversion for S1 binding IgG antibodies | One month after the booster dose
  As measured by ELISA
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies | One month after the booster dose
  As measured by ELISA

SECONDARY OUTCOMES:
Geometric mean fold rise (GMFR) for S1 binding IgG antibodies | One month after the booster dose
  As measured by ELISA
Geometric mean fold rise (GMFR) for S1 binding IgG antibodies in subjects either with or without antibody responses at baseline | One month after the booster dose
  As measured by ELISA
Percentage of participants with seroconversion for S1 binding IgG antibodies in subjects either with or without antibody responses at baseline | One month after the booster dose
  As measured by ELISA
Geometric mean fold rise (GMFR) for SARS-CoV-2 neutralizing antibodies | One month after the booster dose
  As measured by ELISA
Geometric mean fold rise (GMFR) for SARS-CoV-2 neutralizing antibodies in subjects either with or without antibody responses at baseline | One month after the booster dose
  As measured by ELISA
Percentage of participants with seroconversion for SARS-CoV-2 neutralizing antibodies in subjects either with or without antibody responses at baseline | One month after the booster dose
  As measured by ELISA
Change in T-cell IFN-γ secretion from baseline to one month after the booster dose | Baseline and one month after the booster dose
  As measured by IGRA
Incidence of solicited adverse events | For 7 days after the booster dose
  Injection site pain, erythema, swelling, and induration, axillary swelling or tenderness ipsilateral to the side of injection, fever (oral temperature), headache, fatigue, myalgia, arthralgia, nausea, vomiting, and chills, as reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)
Incidence of unsolicited adverse events | For one month after the booster dose
  As reported by the study participants on electronic diaries, and as defined using system organ classes and preferred terms of the Medical Dictionary for Regulatory Activities (MedDRA)

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Nafar, M.D., Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shaheed Labbafinezhad Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No